CLINICAL TRIAL: NCT05675969
Title: Study of Microvesicles in Pre-eclampsia
Brief Title: Pilot Study of Microvesicles in Pre-eclamptic and Non-pre-eclamptic Women With Threatened Preterm Delivery
Acronym: MICROVES-PE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/64
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pre-Eclampsia
Keywords: pre-eclampsia; microvesicles
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A matching will be performed at inclusion between the two groups on gestational age according to two categories: 23-27+6 and 28-31+6 amenorrhoea weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-eclamptic women (Experimental): The intervention consists of the collection of 2 additional tubes of 4.5mL of citrate blood. The sample will be collected as close as possible to the diagnosis of pre-eclampsia during a routine care assessment
  Interventions: Other: Blood sample
- Non pre-eclamptic women (Active Comparator): The intervention consists of the collection of 2 additional tubes of 4.5mL of citrate blood. sampling will be performed during routine care according to the matching.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Collection of 2 additional tubes of 4.5mL of citrate blood

SUMMARY:
A large number of studies on MVs from syncytiotrophoblasts support the hypothesis of their involvement in pre-eclampsia, via their multiple effects, among others as pro-coagulant, immuno-stimulatory and anti-angiogenic factors.

The main objective is to compare the total concentration of the main populations of MVs in the maternal blood of a population of pre-eclamptic patients to those of a population of non-pre-eclamptic patients.

DETAILED DESCRIPTION:
Activated or apoptotic cells release membrane fragments called microvesicles, microparticles, extracellular vesicles or exosomes into the extracellular environment. The term microvesicle (MV) used in this project encompasses all membrane fragments secreted by cells, regardless of their cellular origin, their size or the membrane compartment from which they originate.

The presence on the surface of MVs and in their reservoir of elements from their parent cell, such as surface receptors, mRNAs or microRNAs, led to the hypothesis that MVs could serve as biomarkers, revealing the existence of tissues in distress in the body.

Under physiological conditions, blood plasma contains mainly MVs from red blood cells and platelets, the main circulating cell populations. During pregnancy, the presence of membrane fragments of placental origin in the maternal circulation has long been established. A large number of studies on syncytiotrophoblast-derived MVs support the hypothesis of their involvement in pre-eclampsia, via their multiple effects, among others as pro-coagulant, immuno-stimulatory, anti-angiogenic factors.

The "Membrane Repair and Extracellular Vesicles" team within the CBMN laboratory of the University of Bordeaux has developed original approaches to characterize and quantify MVs, mainly by cryo-electron microscopy, immunogold labeling and flow cytometry. In addition, recent developments from this team allow the analysis of MVs in whole blood, which is a major advantage.

The main objective is to compare the total concentration of the main populations of MVs in the maternal blood of a population of pre-eclamptic patients to those of a population of non-pre-eclamptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Singleton pregnancy (or spontaneously reduced twin pregnancy before 14 SA)
* Gestational age at inclusion between 23 and 31+6 SA
* Collection of the patient's non-opposition
* Affiliated or beneficiary of a social security system
* Specifically for the non-pre-eclampsia group: non-pre-eclamptic patient hospitalized for isolated threat of preterm delivery, whatever the origin, and without clinical (absence of maternal hyperthermia defined by a maternal temperature < 38.0°C) or biological markers of inflammation (CRP<5)
* Specifically for the pre-eclampsia group : diagnosis of severe pre-eclampsia before 32 weeks' gestation

Exclusion Criteria:

* Patient's inability to understand the nature, risks, meaning and implications of the clinical investigation or refusal to give consent
* Patient under legal protection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total concentration of the main MV | baseline
  Total concentration (number of MVs / µL) of the main MV populations, (MVs of erythrocyte, platelet or placental origin, determined by flow cytometry)

SECONDARY OUTCOMES:
Concentration of erythrocyte origin microvesicles | baseline
  Concentration (number of MVs / µL) of MVs of erythrocyte origin by flow cytometry
Concentration of platelet origin microvesicles | baseline
  Concentration (number of MVs / µL) of MVs of platelet origin by flow cytometry
Concentration of placental origin microvesicles | baseline
  Concentration (number of MVs / µL) of MVs of placental origin determined by flow cytometry
Rate of microvesicles | baseline
  Rate of MVs
Number of gravidic hypertension | baseline
  Gravidic hypertension (≥ 160/110 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No